CLINICAL TRIAL: NCT00393250
Title: Hypnosis as a Pain and Symptom Management Strategy in Patients With Sickle Cell Disease
Brief Title: Hypnosis to Manage Pain and Symptoms in Patients With Sickle Cell Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 070011; 07-CC-0011
Record Dates: First submitted 2006-10-26; First posted 2006-10-27 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Sickle Cell Disease; Pain Management
Keywords: Pain Management; Sickle Cell; Sickle Cell Disease; Pain; Hypnosis
MeSH Terms: conditions — Anemia, Sickle Cell; Agnosia; Pain | interventions — Hypnosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1 (Experimental): Hypnosis
  Interventions: Other: Hypnosis
- 2 (Active Comparator): Control
  Interventions: Other: Control

INTERVENTIONS:
Other: Hypnosis — Subjects receive hypnosis (experimental intervention) during 4 weeks of face-to-face encounters with a physician trained in hypnosis. For 6 weeks following the instruction period, the participants will perform daily self- hypnosis using customizable digital media.
  Arms: 1
Other: Control — Subjects in the control arm of the study will receive face-to-face education regarding sickle cell disease for the same length and frequency as the treatment group hypnosis encounters before crossing over to the experimental intervention arm of the study
  Arms: 2

SUMMARY:
This study will examine whether hypnosis can reduce the frequency and intensity of pain in patients with sickle cell disease.

Patients 18 years of age and older with sickle cell disease and a history of pain associated with their disease may be eligible for this study.

Participants are interviewed to assess their frequency and intensity of pain, sleep quality, coping strategies, mood and anxiety and are then randomly assigned to study Group A or B (see below). All participants are given pain diaries to complete at home and turn in at each clinic visit. They undergo the following procedures:

Group A

Weeks 1-4: Receive weekly 60-minute hypnosis sessions, in which they are given suggestions for relieving pain, reducing anxiety, improving sleep and enhancing their health and well-being. The sessions are audio- and videotaped.

Week 5: Are interviewed to assess pain, sleep, coping strategies, mood and anxiety.

Week 6: Receive a DVD player and DVD with instruction on how to perform self-hypnosis. They practice hypnosis at home as often as needed, but at least once a day. They record in a pain diary in the morning and the evening their amount of pain, medication use, school or work attendance, quality and amount of sleep and number of times they use self-hypnosis.

Weeks 8, 10 and 12: Turn in their pain diaries and have a pain assessment.

Week 12: Are assessed for how they respond to the hypnosis.

Group B

Weeks 1-4: Receive weekly 60-minute sessions of education about sickle cell disease.

Week 5: Are interviewed to assess pain, sleep, coping strategies, mood and anxiety.

Week 6: Turn in their daily pain diaries and receive a DVD player and DVD that contains educational materials about sickle cell disease.

Weeks 8, 10 and 12: Turn in their pain diaries and have a pain assessment.

Weeks 13-24: Follow the procedures described in weeks 1-12 for Group A.

DETAILED DESCRIPTION:
Sickle cell disease (SCD) is the most common genetic disease in African-Americans, characterized by recurrent painful vaso-occlusive crises. Standard medical therapies for controlling or preventing crises are limited because of efficacy and/or toxicity. Published studies focus on the frequency of acute pain crises resulting in emergency department use and a number of hospitalizations. However, few studies focus on pain manifestations outside the typical healthcare delivery system. Furthermore, the proportion of patients who are able to self-manage their crises at home without accessing healthcare professionals is unknown. Adjunctive approaches using psychosocial interventions may be effective in further reducing and/or preventing painful crises, as well as in improving quality of life and reducing health care utilization. Recent evidence suggests that learning a cognitive-behavioral intervention centered on self-hypnosis for pain management may be helpful in modulating pain frequency, improving sleep quality, and decreasing use of narcotic pain medications in patients with SCD.

This protocol describes a randomized, controlled, single-crossover, single-blinded pilot study trial of hypnosis for managing pain in SCD patients. Subjects receive hypnosis (experimental intervention) during 4 weeks of face-to-face encounters with a physician trained in hypnosis. For 6 weeks following the instruction period, the participants will perform daily self-hypnosis using customizable digital media. Subjects in the control arm of the study will receive face-to-face education regarding sickle cell disease for the same length and frequency as the treatment group hypnosis encounters before crossing over to the experimental intervention arm of the study. Primary outcome measures include patient assessments of pain frequency, intensity, and quality. Secondary outcome measures include face-to face assessments of psychosocial variables including anxiety, coping strategies, sleep, depression and health-care utilization.

ELIGIBILITY:
* ELIGIBILITY:

Subjects with known or suspected sickle cell disease are eligible to participate in this study.

INCLUSION CRITERIA:

Greater than or equal to 18 years of age.

Diagnosis of Hemoglobin SS sickle cell disease.

Patient identifies history of pain as a significant problem during at least 2 days in the month prior to enrollment.

Written informed consent/assent has been obtained.

<TAB>

EXCLUSION CRITERIA:

Less than 18 years of age.

Unwilling to experience hypnosis or to have hetero-hypnosis sessions recorded.

Non-fluency in written and spoken English.

Physical or other disabilities that prevent adequate participation in hypnotic susceptibility testing.

Does not wish to be video and audiotaped.

Psychosis or psychotic depression.

History of seizures or epilepsy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2007-04-30 (Actual); Primary Completion 2012-06-04 (Actual); Study Completion 2012-06-04 (Actual)

PRIMARY OUTCOMES:
Pain Assessment | 12 weeks
  Pain assessment using 0-10 scale

SECONDARY OUTCOMES:
Face to Face assessment of psychosocial variables | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gwenyth R Wallen, Ph.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (2):
- United States (2):
  - Howard University Hospital, Washington D.C., District of Columbia
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland

REFERENCES:
- [Background] Anbar RD. Self-hypnosis for the treatment of functional abdominal pain in childhood. Clin Pediatr (Phila). 2001 Aug;40(8):447-51. doi: 10.1177/000992280104000804. PMID 11516052
- [Background] Anbar RD. Hypnosis in pediatrics: applications at a pediatric pulmonary center. BMC Pediatr. 2002 Dec 3;2:11. doi: 10.1186/1471-2431-2-11. Epub 2002 Dec 3. PMID 12460456
- [Background] Ballas SK. Sickle cell anaemia: progress in pathogenesis and treatment. Drugs. 2002;62(8):1143-72. doi: 10.2165/00003495-200262080-00003. PMID 12010077
- [Derived] Wallen GR, Middleton KR, Ames N, Brooks AT, Handel D. Randomized trial of hypnosis as a pain and symptom management strategy in adults with sickle cell disease. Integr Med Insights. 2014 Nov 3;9:25-33. doi: 10.4137/IMI.S18355. eCollection 2014. PMID 25520557
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2007-CC-0011.html